CLINICAL TRIAL: NCT04679493
Title: Double Blind, Randomized, Placebo-controlled Study of Safety, Tolerability, and Pharmacokinetics of Ascending Doses of XC7 After Single and Multiple Oral Administration in Healthy Volunteers
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics of XC7 (Which is Planned Use in the Treatment of COVID-19) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NP Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-XC7-01
Record Dates: First submitted 2020-12-18; First posted 2020-12-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Healthy Volunteers
Keywords: Coronavirus; Phase I
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: The dose cohorts cohorts will be included into the study subsequently based on preliminary safety results evaluation performed by the DSMC. 2 doses of XC7/placebo (100 mg, 200 mg) were used in the study.The duration of exposure to the ID is planned 1 day in single dosing cohorts and 14 days in multiple dosing cohort.
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using placebo equivalent to XC7 capsules without active pharmaceutical ingredients (API) and the corresponding labeling of the ID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- XC7 100 mg single (Experimental): Cohort 1 - 4 subjects will be randomized in a 3:1 ratio to be treated either XC7 100 mg (3 subjects) or placebo (1 subject, see placebo single arm)
  Interventions: Drug: XC7 100 mg single
- XC7 200 mg single (Experimental): Cohort 2 - 4 subjects will be randomized in a 3:1 ratio to be treated either XC7 200 mg (3 subjects) or placebo (1 subject, see placebo single arm)
  Interventions: Drug: XC7 200 mg single
- Placebo single (Placebo Comparator): Placebo comparator arm will consist of 2 subjects (1 subject from Сohorts 1 and 2)
  Interventions: Drug: Placebo single
- XC7 200 mg multiple (Experimental): Cohort 3 - 6 subjects will be randomized in a 6:2 ratio to be treated either XC7 200 mg (6 subjects) or placebo (1 subject, see placebo multiple arm)
  Interventions: Drug: XC7 200 mg multiple
- Placebo multiple (Placebo Comparator): Placebo comparator arm will consist of 2 subjects from cohort 3
  Interventions: Drug: Placebo multiple

INTERVENTIONS:
Drug: XC7 100 mg single — The volunteers will receive a single dose of the ID (1 capsule once, 100 mg)
  Arms: XC7 100 mg single
Drug: XC7 200 mg single — The volunteers will receive a single dose of the ID (2 capsules once, 100 mg each)
  Arms: XC7 200 mg single
Drug: Placebo single — The volunteers will receive a single dose of the ID (1 or 2 capsules once)
  Arms: Placebo single
Drug: XC7 200 mg multiple — The volunteers will receive multiple doses of the ID during 14 days (2 capsules daily, 100 mg each)
  Arms: XC7 200 mg multiple
Drug: Placebo multiple — The volunteers will receive multiple doses of the ID during 14 days (2 capsules daily)
  Arms: Placebo multiple

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety, tolerability and pharmacokinetics (PK) of ascending doses of XC7 after single and multiple oral administration in healthy volunteers. It's planned to include sequentially 2 cohorts of 4 volunteers who will receive a single dose of XC7 (100 mg and 200 mg) or placebo (cohort ratio 3:1) and 1 cohort of 8 volunteers who will receive multiple doses of the XC7 (200 mg) or placebo during 14 days (cohort ratio 6:2).

DETAILED DESCRIPTION:
The study will be conducted in 1 centre. The study will consist of 3 periods: screening (7 days), treatment (1 or 14 days) and follow-up (7 or 28 days).

The volunteers of single dosing cohorts will receive the investigated drug (ID) ХС7 or placebo once and stay at the study center for at least 24 hours after the ID administration to monitor the safety parameters and for sampling for PK analysis. The Follow-up will last 7 days, during which safety parameters and PK in volunteers will be studied. Based on all safety data from the XC7 100 mg cohort, the Data Safety Monitoring Committee (DSMC) will consider dose increase and entry of the 200 mg cohort. If the single dose of ХС7 200 mg is considered to be safe, the third multiple dosing cohort of 200 mg will be included in the study.

The volunteers from multiple dosing cohort will receive the ID (ХС7 or placebo) once a day during 14 days and will stay at the hospital (study center) during the first five days after administration of the ID. The Follow-up will last 14 days, during which they will study safety parameters and PK in volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking men (nonsmokers at least within the last year before the screening) at the ages from 18 through 45;
2. Verified diagnosis "healthy" according to standard clinical, laboratory and instrumental methods of examination;
3. Body mass index from 18.5 to 30.0 kg/m2 with body weight of more than 45 kg and no more than 110 kg;
4. Negative result for alcohol vapor content in the exhaled air, narcotic substances in the urine;
5. Agreement to use adequate contraception methods during the study and 3 months after its completion: condoms with spermicide (foam, gel, cream, suppository);
6. Signed patient explanation sheet and informed consent for participation in the study.

Exclusion Criteria:

1. Chronic diseases of the cardiovascular, bronchopulmonary, nervous, endocrine, musculoskeletal system, as well as the gastrointestinal tract, liver, kidneys, blood, mental illness, epilepsy or convulsive seizures;
2. Abnormal results of standard laboratory tests and investigations at the screening visit;
3. Gastrointestinal surgery (except for appendectomy) in the past medical history;
4. Systolic blood pressure of less than 90 mm Hg or above 139 mm Hg, diastolic blood pressure of less than 60 mm Hg or above 90 mm Hg, heart rate of less than 60 bpm or above 90 bpm - at screening;
5. Regular administration of drugs within 2 weeks prior to screening (including herbal agents and dietary supplements);
6. Use of drugs with significant effect on hemodynamics, hepatic function, etc. (e.g. barbiturates, omeprazole, cimetidine, etc.) within 30 days prior to screening;
7. Antibodies to HIV and hepatitis C, hepatitis B surface antigen, positive test for syphilis;
8. Unstable sleep architecture (e.g. night work, sleep disorders, insomnia, recently returned from another time zone, etc.), extreme physical activity (e.g. weight lifting);
9. Special diet (for example, vegetarian, vegan, low calorie (less than 1000 kcal/day));
10. Signs of alcohol abuse (intake of more than 10 units of alcohol per week) or 50 ml of hard alcohol; drinking alcohol within 4 days prior to screening;
11. Signs of drug abuse; taking narcotic and psychotropic drugs (opiates/morphine, methamphetamine, amphetamine, cannabinoids/marijuana, cocaine, methadone, ecstasy, tricyclic antidepressants, barbiturates) at the moment and in the history;
12. burdened past allergic history;
13. Hypersensitivity to the components of the investigated drugs;
14. Blood/plasma donation (from 450 ml blood or plasma) within 2 months prior to screening;
15. Participation in other clinical studies within 3 months prior to screening;
16. Acute infectious diseases within 4 weeks prior to screening;
17. Inability to read or write; unwillingness to understand and follow the procedures of the study protocol; noncompliance with the drugs administration or procedures schedule, which according to the researchers may affect the study results or the volunteer safety and prevent the further participation of the volunteer in the study; any other associated medical or serious mental conditions that make the volunteer inadequate for participation in the clinical study and restrict the validity of informed consent or may affect the volunteer's ability to participate in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events (AEs) per treatment arm | Day -7 (7 days before first dose) - Day 58
  Adverse events will be classified according to CTCAE ver 4.03. Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version.

SECONDARY OUTCOMES:
Pharmacokinetics of XC7 by assessing AUC0-inf | Day 1 - Day 4
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity.
Pharmacokinetics of XC7 by assessing Cmax | Day 1 - Day 4
  Maximum plasma concentration
Pharmacokinetics of XC7 by assessing AUC0-t | Day 1 - Day 4
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of XC7 by assessing Tmax | Day 1 - Day 4
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of XC7 by assessing T1/2 | Day 1 - Day 4
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Autonomous Educational Institution of Higher Education "The First Moscow State Medical University named after I.M. Sechenov" of the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No